CLINICAL TRIAL: NCT05659433
Title: Contrast-enhanced vs. B-mode Ultrasound-guided Percutaneous Biopsy of Retroperitoneal Tumors - a Randomized Controlled Trial
Brief Title: Contrast-enhanced vs. B-mode Ultrasound-guided Percutaneous Biopsy of Retroperitoneal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Principal Investigator, Rareș Crăciun, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CEUS-PBRT
Record Dates: First submitted 2022-12-03; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Retroperitoneal Neoplasms
Keywords: Percutaneous biopsy; Contrast-enhanced ultrasonography; CEUS; Retroperitoneal neoplasms
MeSH Terms: conditions — Retroperitoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-mode Ultrasound-guided Biopsy (Active Comparator)
  Interventions: Procedure: B-mode US-guided percutaneous biopsy
- Contrast-enhanced Ultrasound-guided Biopsy (Experimental)
  Interventions: Procedure: CEUS-guided percutaneous biopsy

INTERVENTIONS:
Procedure: CEUS-guided percutaneous biopsy — A standard dose of SonoVue ultrasound contrast agent is injected prior to the biopsy, and the percutaneous biopsy is guided in real time, targeting the contrast-enhanced areas of the retroperitoneal tumors (viable, vascularized)
  Arms: Contrast-enhanced Ultrasound-guided Biopsy
Procedure: B-mode US-guided percutaneous biopsy — Standard of care (B-mode) ultrasound-guided percutaneous biopsy, without contrast enhancement
  Arms: B-mode Ultrasound-guided Biopsy

SUMMARY:
Background: Retroperitoneal tumors are typically large and inhomogeneous, with a variable amount of necrosis within the tumor mass which decreases the diagnostic yield of biopsy (false negative or inadequate).

Rationale: Real-time contrast enhancement can highlight the viable tumoral tissue and avoid the necrotic area.

Aims: To compare contrast-enhanced ultrasound (CEUS) guidance and conventional (B-mode) ultrasound (US) guidance in terms of diagnostic yield, need for repeat biopsy, and rate of adverse events.

Methods: A consecutive series of patients with previously documented retroperitoneal tumors and indications for percutaneous biopsy were randomly assigned to benefit from the standard of practice B-mode US-guided biopsy or CEUS-guided biopsy.

The diagnostic accuracy, need for repeat biopsy, and adverse events were noted.

ELIGIBILITY:
Inclusion Criteria:

* All patients with retroperitoneal tumors with indication for percutaneous biopsy

Exclusion Criteria:

* Tumors inaccessible for ultrasound guided biopsy
* Standard contraindications for biopsy (altered coagulation tests, poor performance status)
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with a biopsy sample adequate for pathology interpretation | 4 weeks

SECONDARY OUTCOMES:
Number of patients requiring a second biopsy due to prior inadequate sampling | 6 weeks
Number of patients with procedural-related adverse events | One week
  Bleeding, hematoma, puncture-site infection, prolonged hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Spârchez, MD, Prof., Study Chair — Prof. Dr. O. Fodor Regional Institute of Gastroenterology and Hepatology, Cluj-Napoca
Locations (1):
- Prof. Dr. O. Fodor Regional Institute of Gastroenterology and Hepatology, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No